CLINICAL TRIAL: NCT04003194
Title: Impact of Pinto Beans as Part of a Normal Diet on Glycemic Control in Adults With Type 2 Diabetes: a Randomized Trial
Brief Title: Pinto Beans and Glycemic Control in Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Collaborators: Iowa State University (Other)
Responsible Party: Principal Investigator, Andrea Hutchins, Associate Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UCCS09-028
Record Dates: First submitted 2019-06-24; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes
Keywords: pulses; legumes; Phaseolus vulgaris L.; glycemic response
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Crossover design with 2-12 week intervention and comparator phases separated by a 4-week washout.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pinto beans (Experimental): 1/2 cup pinto beans eaten daily by free-living individuals for 12 consecutive weeks.
  Interventions: Other: Pinto Beans
- Green beans (Active Comparator): 1/2 cup green beans eaten daily by free-living individuals for 12 consecutive weeks.
  Interventions: Other: Green Beans - control

INTERVENTIONS:
Other: Pinto Beans — The intervention was 1/2 cup of pinto beans each day.
  Other Names: Pinto Beans - intervention
  Arms: Pinto beans
Other: Green Beans - control — The control was 1/2 cup of green beans each day.
  Other Names: Control
  Arms: Green beans

SUMMARY:
This study examines the impact of daily consumption of ½ c pinto beans, compared to a control (½ c green beans), on fasting glucose, postprandial glucose and HbA1c concentrations in adults with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This study utilized a randomized, pretest-posttest, crossover (within-group) design, that includes two treatment periods [control period (½ c. green beans each day) and pinto beans (½ c each day)], each 12-weeks in duration with a 4- week wash-out period to determine the impact on fasting glucose, postprandial glucose and HbA1c concentrations. After a baseline wash-in period, 16 participants are randomly assigned to 2 treatment periods [control period and pinto beans], each 12-weeks in duration. On 28 randomized days during the wash-in period and interventions, participants keep diet records and measure a postprandial capillary glucose concentration using a glucometer 1 hour after the meal during which the pinto beans or control are consumed. Before and after each 12-week intervention, participants provide a fasted venous blood sample for glucose and HbA1c analyses.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of T2DM by a physician;
* currently attempting control of T2DM by diet or metformin;
* fasting glucose ≥ 90 mg/dL (confirmed by fasting blood draw or potential participant provided lab analysis conducted within last 30 days) and/or hemoglobin A1C ≥ 6.5% (confirmed by blood draw or potential participant provided lab analysis conducted within last 30 days);
* body mass index (BMI) of 22-40 kg/m2;
* no unresolved health conditions and no diagnosis of gastrointestinal disease;
* limited history of legume intake;
* willingness to follow study protocol, scheduling, and ability to come to the testing location;
* no recent weight gain or loss (>10% over 6 months);
* no use of medications and/or dietary supplements other than metformin that affected glucose;
* women could not be pregnant or breastfeeding;
* habitual alcohol consumption had to be less than 2 drinks per day (specifically ≤ 720 ml of beer, 240 ml of wine, or 90 ml of hard liquor).

Exclusion Criteria:

* Non compliance with above inclusion criteria.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Glucose | 12 weeks pre and post
  Change in fasting blood glucose levels

SECONDARY OUTCOMES:
Postprandial glucose | 1 time per week from week 1 of each intervention to week 12 of each intervention
  1 time per week from week 1 of each intervention to week 12 of each intervention
Change in Hemoglobin A1c | 12 weeks pre and post
  Change in Blood hemoglobin A1c

IPD SHARING:
Plan to Share IPD: No